CLINICAL TRIAL: NCT03236584
Title: Investigation of Efficacy of Tenofovir Monotherapy in Comparison With Lamivudine Plus Adefovir in Patients With Chronic Hepatitis B Patients Who Had Achieved Complete Viral Suppression on Lamivudine Plus Adefovir Combination Therapy - Multicenter Randomized Open-label Controlled Trial
Brief Title: Tenofovir Monotherapy in Patients With Chronic Hepatitis B Patients Who Had Achieved Complete Viral Suppression on Lamivudine Plus Adefovir
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Uijeongbu St. Mary Hospital (Other)
Responsible Party: Principal Investigator, Chang Wook Kim, C.W. Kim, Uijeongbu St. Mary Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UC15MISI0099
Record Dates: First submitted 2017-07-28; First posted 2017-08-02 (Actual); Last update posted 2017-08-02 (Actual); Status verified 2017-07

CONDITIONS: Proportion of Patients With a Sustained Virological Response (Serum HBV DNA <20 IU/mL) at Week 48
MeSH Terms: interventions — Lamivudine; Tenofovir

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- lamivudine adefovir (Active Comparator)
  Interventions: Drug: lamivudine plus adefovir combination
- tenofovir (Experimental)
  Interventions: Drug: Tenofovir Disoproxil Fumarate

INTERVENTIONS:
Drug: lamivudine plus adefovir combination — continuing lamivudine plus adefovir
  Arms: lamivudine adefovir
Drug: Tenofovir Disoproxil Fumarate — switching to tenofovir
  Arms: tenofovir

SUMMARY:
Little is known about efficacy of switching to tenofovir monotherapy for lam-resistant chronic hepatitis B patients who achieved a complete virological response to lamivudine plus adefovir. This study was to investigate the efficacy of switching to tenofovir monotherapy for lamivudine -resistant chronic hepatitis B patients with undetectable hepatitis B virus DNA while on lamivudine plus adefovir combination therapy

ELIGIBILITY:
Inclusion Criteria:

* HBsAg (+) for > 6 months age >19 years antiviral resistance to LAM (rtL180M and/or M204V/I) currently receiving LAM plus ADV for more than 12 months HBV DNA levels <20 IU/ml on two consecutive tests of 3-month interval

Exclusion Criteria:

* Cr ≥1.5 mg/dL Evidence of decompensated liver disease Malignant neoplasm Coinfection with HIV, HCV

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2018-03-30 (Estimated); Study Completion 2019-03-30 (Estimated)

PRIMARY OUTCOMES:
SVR | 48 WEEK
  Proportion of patients with a sustained virological response (serum HBV DNA <20 IU/mL) at week 48

IPD SHARING:
Plan to Share IPD: No